CLINICAL TRIAL: NCT00788632
Title: Improving Care of Osteoporosis: Multi-Modal Intervention to Increase Testing and Treatment (ICOMMIITT)
Acronym: ICOMMIITT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: Kaiser Permanente (Other)
Responsible Party: Principal Investigator, Kenneth Saag, MD, MSc, Professor of Medicine, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: X080219004
Record Dates: First submitted 2008-11-07; First posted 2008-11-11 (Estimated); Last update posted 2013-03-22 (Estimated); Status verified 2013-03

CONDITIONS: Osteoporosis
Keywords: Osteoporosis; BMD; Bisphosphonates; Educational materials; Patient Stories
MeSH Terms: conditions — Osteoporosis | interventions — Drug Delivery Systems

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- educational materials (Experimental): Patient educational DVD and brochure
  Interventions: Behavioral: Patient educational DVD and brochure
- physician education (Other): Physician web modules
  Interventions: Behavioral: Physician web modules
- System intervention (Experimental): Self-referral letter with toll-free number provided
  Interventions: Behavioral: System

INTERVENTIONS:
Behavioral: Patient educational DVD and brochure — Construct a tailored direct-to-patient intervention to educate and activate older women about osteoporosis testing and treatment and aimed at improving patient-provider communication and "closing the loop" between knowledge communication and action. The intervention will include risk assessment, will be delivered through culturally/ethnically tailored "story-telling", and will be mailed-out as both a paper copy (Booklet) and an interactive DVD (allowing the patient to use the delivery mediums they are most comfortable with). A follow-up brochure will be sent as a "booster".
  Arms: educational materials
Behavioral: Physician web modules — Web based osteoporosis continuing medical education (CME) materials
  Arms: physician education
Behavioral: System — Create a practice redesign strategy to alert patients that they should receive a BMD test and provide them with direct patient access to schedule their own test
  Arms: System intervention

SUMMARY:
The purpose of this study is to rigorously test the incremental impact of simple, generalizable interventions to improve healthcare among older women at high risk for osteoporosis. Building on the experience of our University of Alabama at Birmingham (UAB) interdisciplinary team we have designed an innovative, scientifically rigorous, and highly feasible implementation research project in partnership with two Kaiser Permanente (KP) research centers. Kaiser Permanente, one of the Nation's largest Healthcare Organizations, uses an integrated electronic medical record (EMR), with full capture of pharmacy, clinical (including BMD results), and claims data, and cares for a racially/ethnically, socio-economically, and geographically diverse population. To address innovative questions in implementation research, we will perform a multi-modal group randomized trial involving over 18,000 patients seen by over 330 primary care providers (PCPs) at 25 KP facilities in the Northwest and Southeast. If proven effective, our system-centered and patient-centered approach will advance the state of implementation science and be applicable to evidence implementation in other musculoskeletal disorders and to other health care settings.

ELIGIBILITY:
Inclusion Criteria:

* female
* age 65 or older

Exclusion Criteria:

* prior osteoporosis testing (BMD)
* prior osteoporosis treatment

Min Age: 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 12128 (Actual)
Dates: Start 2010-05; Primary Completion 2011-12 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Bone Mineral Density (BMD) testing | 12 months

SECONDARY OUTCOMES:
Osteoporosis prescription medications | 12 months
Patient-Physician communication regarding osteoporosis treatment and testing | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth G Saag, MD, MSc, Principal Investigator — University of Alabama at Birmingham
Locations (2):
- United States (2):
  - Kaiser Permanente Southeast, Atlanta, Georgia
  - Kasier Permanente Northwest, Portland, Oregon